CLINICAL TRIAL: NCT05433857
Title: Evaluation of the Clinical Outcome of Probiotics in Systemic Lupus Erythematosus
Brief Title: Probiotics in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Sayed Fouad, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC 80
Record Dates: First submitted 2022-06-17; First posted 2022-06-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Probiotics; Lactobacillus; Systemic lupus erythematosus; SLEDAI-2K
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Interventional, Prospective, randomized, controlled, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 20 patients will receive the standard therapy for 12 weeks
- Interventional group (Experimental): 20 patients will receive the standard therapy in addition to two capsules once daily of probiotic Lacteol Forte® Capsules for 12 weeks
  Interventions: Drug: Lacteol forte capsules

INTERVENTIONS:
Drug: Lacteol forte capsules — probiotic Lacteol Forte® capsules (5 billion heat-killed Lactobacillus LB, corresponding to lactobacillus delbruekii and lactobacillus fermentum) Two capsules are To be taken once daily
  Other Names: lactobacillus delbruekii and lactobacillus fermentum
  Arms: Interventional group

SUMMARY:
Dysbiosis, or disruption of the gut microbiota, leads to the onset of autoimmunity. Increasing data suggest that the gut microbiota is changed in various murine lupus models as well as in human systemic lupus erythematosus SLE patients. Ingestion of lactobacilli, which have immunoregulatory properties, may be a viable strategy for controlling disease development and progression in patients with lupus, such as increasing the remission period and decreasing flare frequency.

DETAILED DESCRIPTION:
1. Patients will be recruited and evaluated for eligibility.
2. Patients who met the eligibility criteria will be randomly assigned to either control or interventional group.
3. Patients in the control group will receive their standard therapy for 12 weeks and patients in the interventional group will receive their standard therapy plus one sachet daily of lacteol forte sachets for 12 weeks.
4. Collection of demographic data, full medication history, and full medical history will be performed at baseline and every 4 weeks.
5. Assessment of disease activity using SLEDAI-2K score, quality of life using the validated Arabic LupusPROv1.8 questionnaire, and Pain assessment using the validated Arabic version of the Short-Form McGill Pain Questionnaire will be performed at baseline and at the end of the study.
6. Safety and tolerability monitoring will be performed weekly using a side effect and/or adverse effect monitoring sheet.
7. Blood and urine samples for laboratory investigations will be withdrawn at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years, male or female.
2. Patients are willing to sign a written informed consent.
3. Patients fulfilling American college of rheumatology classification criteria for SLE.
4. Patients diagnosed with active systemic lupus erythematosus defined as SLEDAI-2K score more than 4.

Exclusion Criteria:

1. Patients ˂ 18 years or ˃65 years of age.
2. Patients with a history of drug allergies to probiotics administration.
3. Pregnant or breastfeeding females.
4. Current probiotics use.
5. Patients scheduled for surgical intervention during the study period or up to 2 weeks after the end of the study.
6. patients suffering from active severe neuropsychiatric manifestations of SLE.
7. Patients with other auto-immune diseases.
8. Patients suffering from any type of cancer.
9. patients participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | At baseline and at 12 weeks
  Change in disease activity measured by SLEDAI-2K score. The most appropriate SLEDAI-2K cut-off score for definition of active disease which links to the need to increase therapy is 3 or 4

SECONDARY OUTCOMES:
Improvement of immunologic parameters | At baseline and at 12 weeks
  Anti-dsDNA levels
Improvement of serum complement | At baseline and at 12 weeks
  Complements 3 and 4
patients' quality of life | At baseline and at 12 weeks
  Assessment of patients' quality of life using the validated Arabic Lupus Patient-reported outcome survey version 1.8 (LupusPROv1.8)
Pain assessment | At baseline and at 12 weeks
  Pain assessment using the validated Arabic version of the Short-Form McGill Pain Questionnaire
Incidence of potential adverse effects | Weekly up to 12 weeks
  Monitoring for side and/or adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Rana Sayed, PhD, Study Director — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasseya, Egypt

IPD SHARING:
Plan to Share IPD: No